

# Assessing the safety of discontinuing non-selective beta-blockers in cirrhotic patients with managed primary aetiological factors according to Baveno VII consensus

(Short title: Stop-NSBB Study)

#### **Clinical study protocol**

Prepared by:

Vincent Wong

Professor

Department of Medicine and Therapeutics

The Chinese University of Hong Kong

Version 1.0

Date: 4 Dec 2023

### Table of Contents

| 1. B | ACKGROUND | 3 |
|---|---|---|
| 1.1 | Significance of cirrhosis and portal hypertension | 3 |
| 1.2 | Non-invasive assessment of portal hypertension | 3 |
| 1.3 | Emerging concept: hepatic recompensation and reversal of cirrhos 4 | sis and portal hypertension |
| 2. S' | TUDY OBJECTIVES | 4 |
| 3. S | TUDY DESIGN OVERVIEW | 4 |
| 4. P | ATIENTS | 5 |
| 4.1 | Inclusion criteria | 5 |
| 4.2 | Exclusion criteria | 5 |
| 5. C | CLINIC VISITS AND ASSESSMENTS | 6 |
| 5.1 | Clinical assessments | 6 |
| 5.2 | Vibration-controlled transient elastography | 6 |
| 5.3 | Upper gastrointestinal endoscopy | 7 |
| 5.4 | Follow-up | 7 |
| 6. D | DATA PROCESSING AND ANALYSIS | 7 |
| 6.1 | Analysis datasets | 7 |
| 6.2 | Primary endpoint | 8 |
| 6.3 | Secondary endpoints | 8 |
| 6.4 | Sample size calculation | 9 |
| 6.5 | Anticipated challenges and contingency plans | 9 |
| 7. E | THICS | 10 |
| 7.1 | Ethics review | 10 |
| 7.2 | Ethical conduct of the study | 10 |
| 7.3 | Informed consent | 10 |
| 7.4 | Data sharing | 11 |
| 8. A | ADVERSE EVENT REPORTING | 11 |
| 8.1 | Adverse events | 11 |
| 8.2 | Serious adverse events | 12 |
| 9 RFF | FERENCES | 12 |

#### 1. BACKGROUND

#### 1.1 Significance of cirrhosis and portal hypertension

Liver cirrhosis is the common final pathway of various chronic liver diseases. Globally, mortality due to cirrhosis have risen from 899 000 in 1990 to 1.32 million deaths in 2017. Additionally, as of 2017, 112 million and 10.6 million people were living with compensated and decompensated cirrhosis, respectively (1). Portal hypertension stands out as the primary cause of cirrhotic complications, such as ascites and variceal haemorrhage. Accurate diagnosis of clinically significant portal hypertension is crucial because the administration of non-selective beta-blockers (NSBBs) can reduce the risk of variceal haemorrhage and hepatic decompensation (2, 3).

Chronic liver disease is highly prevalent in Hong Kong. A community screening study in Hong Kong in 2015-2016 indicated that the prevalence of hepatitis B surface antigen was still 7.8% (4). Studies by our group have further highlighted the extent of the problem, revealing that 26% of the local population and a staggering 73% of patients with type 2 diabetes suffer from metabolic dysfunction-associated steatotic liver disease (5, 6). These chronic liver diseases carry a significant risk of progressing to cirrhosis and hepatic decompensation.

#### 1.2 Non-invasive assessment of portal hypertension

Historically, the gold standard for assessing portal hypertension requires the measurement of hepatic venous pressure gradient, an invasive procedure rarely performed outside research settings (7). However, accumulating data support the use of non-invasive tests to assess portal hypertension. Specifically, liver stiffness measurement (LSM) through vibration-controlled transient elastography reflects the degree of liver fibrosis and the severity of cirrhosis. Furthermore, the platelet count reflects whether a patient with cirrhosis has hypersplenism secondary to portal hypertension. Additionally, spleen stiffness measurement (SSM) may be an even more direct evaluation of portal hypertension and has been used to ascertain improvements in portal hypertension following the initiation of NSBB (8, 9). Based on existing data, the latest Baveno VII consensus has endorsed the use of these non-invasive tests to rule out (if LSM <15 kPa and platelet count >150×10<sup>9</sup>/L) and to confirm (if LSM ≥25 kPa) the presence of clinically significant portal hypertension (10).

In a randomised controlled trial involving 548 patients with radiological cirrhosis, our group demonstrated that LSM+SSM was non-inferior to routine endoscopy in detecting varices and preventing future variceal haemorrhage (11, 12). Furthermore, we validated the use of LSM-based criteria for excluding the presence of varices requiring treatment across a range of chronic liver diseases, including patients with or without hepatocellular carcinoma (13-15). Additionally, we reported the natural history of patients falling within the grey zone according to the Baveno VII criteria. Importantly, we identified factors associated with hepatic decompensation in this specific patient population (16).

## 1.3 Emerging concept: hepatic recompensation and reversal of cirrhosis and portal hypertension

As a number of chronic liver diseases can now be well controlled or cured, it is increasingly apparent that cirrhosis can resolve over time when the primary aetiology is controlled (17). Reports have also emerged, suggesting an improvement in portal hypertension and even hepatic recompensation in such circumstances (18). This has led to the practical recommendation on discontinuing NSBB in patients with LSM <25 kPa after removal or suppression of the primary aetiological factor, in the absence of varices (10). Removal or suppression of the primary aetiological factor includes sustained virological response in chronic hepatitis C, complete hepatitis B virus DNA suppression in chronic hepatitis B patients, and long-term abstinence from alcohol in those with alcohol-related liver disease. Nonetheless, it is crucial to note that these recommendations are based on tenuous evidence (C.2 recommendation). While cessation of NSBB in patients no longer requiring it can reduce unnecessary expenses (prescription and monitoring) and side effects, it remains imperative to confirm the safety of this approach through well-designed, prospective studies.

#### 2. STUDY OBJECTIVES

- 1. We aim to test the hypothesis that recurrent varices will occur in less than 5% of patients with cirrhosis who discontinue non-selective beta-blockers (NSBBs) in accordance with the Baveno VII consensus (i.e., effective management or removal of primary aetiological factor, liver stiffness measurements below 25 kPa, and absence of varices confirmed by endoscopy).
- 2. We aim to assess the hypothesis that variceal haemorrhage will occur in less than 5% patients with cirrhosis who cease NSBB use, adhering to the Baveno VII guidelines.
- 3. We aim to identify factors associated with recurrent varices and variceal haemorrhage, with a special focus on serial liver and spleen stiffness measurements obtained by vibration-controlled transient elastography.

#### 3. STUDY DESIGN OVERVIEW

This study is designed as a multicentre, prospective cohort investigation. The study consists of three main parts:

Part 1: We will perform endoscopy on patients with LSM <25 kPa. This part aims to identify both the percentage of patients harbouring varices and the factors associated with their presence.

**Part 2:** Patients without varices will discontinue NSBB and undergo prospective follow-up. Endoscopy will be repeated at 1 year to determine the rate of recurrent varices and any contributing factors.

**Part 3**: Patients will continue prospective follow-up to determine the incidence and factors associated with hepatic decompensation, including variceal haemorrhage, with prespecified outcome analysis at 3- and 10-year marks.

Although the study's follow-up extends beyond the financial coverage of the General Research Fund, patients will still continue at least annual follow-up at the participating centres as part of the standard care, with endpoints ascertained at each visit. The General Research Fund will finance Parts 1 and 2 of this project and establish a valuable cohort for the collection of outcome data.

#### 4. PATIENTS

Eligible patients will be identified from the general medical and hepatology clinics in Hong Kong and collaborating countries. At present, investigators from France, Singapore and Malaysia have confirmed their participation.

#### 4.1 Inclusion criteria

To be eligible for enrolment, patients must meet all the following criteria:

- Aged 18 years or above
- Evidence of cirrhosis, based on either radiological and/or clinical features
- History of varices, variceal haemorrhage or portal hypertension warranting NSBB
- Removal or suppression of the primary aetiological factor (i.e., sustained virological response in chronic hepatitis C, complete hepatitis B virus DNA suppression in chronic hepatitis B, and long-term alcohol abstinence in alcohol-related liver disease)
- LSM <25 kPa
- Provision of written informed consent

#### 4.2 Exclusion criteria

Patients with any of the following will be excluded from the study:

- Active aetiological factors not addressed in the inclusion criteria (e.g., autoimmune or hereditary liver diseases). However, hepatic steatosis—commonly coexisting with other liver diseases—is not an exclusion criterion unless accompanied by high plasma alanine aminotransferase >40 U/L or confirmed steatohepatitis.
- Recent hepatic decompensation within the past year (total bilirubin >50 μmol/L, prothrombin time >1.3 times the upper normal limit [unless attributable to use of anti-coagulation], albumin <35 g/L, or presence of ascites, variceal haemorrhage or hepatic encephalopathy). Notably, the Baveno VI criteria used LSM <20-25 kPa and normal platelet count >150×10<sup>9</sup>/L to rule out varices requiring

treatment (19). However, in line with the Baveno VII consensus, which sets an LSM <25 kPa as the threshold for considering NSBB discontinuation, thrombocytopenia is not an exclusion criterion to allow the cohort to include a wider spectrum of patients.

- Current or history of hepatocellular carcinoma.
- Radiological evidence of portal vein thrombosis.
- History of other malignancies (unless in complete remission for >5 years).
- History of liver transplantation or liver resection.
- Contraindications to undergoing endoscopy.
- Other clinical indications for NSBB (e.g., cardiovascular disease, arterial hypertension)

#### 5. CLINIC VISITS AND ASSESSMENTS

#### 5.1 Clinical assessments

The following procedures will be performed at baseline, month 3, month 6, and year 1:

- Documentation of medical history and new symptoms
- Documentation of hepatic events and their dates of occurrence (i.e., ascites, spontaneous bacterial
  peritonitis, variceal haemorrhage, hepatic encephalopathy, hepatorenal syndrome-acute kidney
  injury, hepatocellular carcinoma, liver transplantation; detailed definitions provided in the full
  protocol)
- Dates and causes of death for patients who pass away between visits will be recorded
- Standard questionnaires will be used to document smoking and alcohol consumption
- Physical examination
- Anthropometric measurements including body weight, height, waist and hip circumferences, will be collected. Body mass index will be calculated as body weight (kg) divided by height (m) squared
- Blood pressure and pulse rate measured after a 15-minute rest
- Blood tests will include complete blood count, prothrombin time, renal function test, liver blood test (including alanine aminotransferase, aspartate aminotransferase and gamma-glutamyl transpeptidase), and alpha-fetoprotein
- Store 10 mL of clotted blood and 10 mL of EDTA blood for future genetic and biochemical research (with separate consent)

#### 5.2 Vibration-controlled transient elastography

LSM and SSM assessments will be carried out using vibration-controlled transient elastography (FibroScan 630 Expert, Echosens, Paris, France). Operators with a minimum of 500 examinations completed and trained according to the manufacturer's guidelines will conduct the tests (20). Examinations will be performed at baseline, month 3, month 6, and year 1. Ten measurements will be

recorded each for the liver and spleen, and their median value will be used to derive the corresponding stiffness. The machine's automated probe selection tool will determine the use of M and XL probes for LSM, while the dedicated 100Hz probe will be required for SSM.

LSM is considered reliable if there are ten or more valid measurements, and the interquartile range-to-median ratio of the measurements is  $\leq 0.3$ . While no standardised reliability criteria exist for SSM, variability of SSM will be tracked in this study.

#### 5.3 Upper gastrointestinal endoscopy

Upper gastrointestinal endoscopy will be performed by experienced endoscopists with a minimum of 100 prior examinations, at baseline and year 1. The scope of the examination will include the oesophagus, stomach, and the first and second parts of the duodenum. The size of varices will be graded using the modified Paquet classification (grade I for varices extending just above the mucosal level; grade II for varices projecting by one-third of the luminal diameter and non-compressible upon air insufflation; and grade III for varices projecting up to 50% of the luminal diameter and in contact with each other) (21). Additionally, the location and presence of red wale markings and cherry red spots will be documented.

#### 5.4 Follow-up

Other follow-up procedures will be considered part of the standard of care and will be covered by local resources. These include but are not limited to the treatment of chronic liver disease and co-morbid conditions as well as surveillance for hepatocellular carcinoma through periodic abdominal ultrasonography and/or alpha-fetoprotein testing. Patients will be scheduled for at least one annual visit or more frequently, as clinically indicated. At each visit, incident hepatic events will be documented.

#### 6. DATA PROCESSING AND ANALYSIS

#### 6.1 Analysis datasets

**Part 1:** This analysis will include all eligible patients who meet the inclusion and exclusion criteria and undergo endoscopy at baseline.

**Part 2**: The intention-to-treat analysis will include all patients with no varices at baseline and have discontinued at least one dose of NSBB. Those who resume NSBB or are lost to follow-up will be classified as treatment failures (i.e., assumed to have recurrent varices). The per- protocol analysis will focus on all patients who undergo follow-up endoscopy at 1 year or resume NSBB, with the resumption of NSBB being classified as treatment failure, as previously noted.

**Part 3**: This part will include all patients with no varices at baseline who have also discontinued at least one dose of NSBB. Data will be censored at the point of patient death or liver transplantation. Patients who experience relapses of the primary aetiological factor (e.g., recurrent hepatitis C virus infection, virological breakthrough in chronic hepatitis B, and relapse of alcohol consumption) will be given the options to either resume NSBB or continue regular surveillance by transient elastography according to the Bayeno VI criteria.

#### 6.2 Primary endpoint

The primary endpoint of this study is recurrent varices at the one-year mark among patients who have discontinued NSBB. Due to substantial intra- and inter-observer variability in the diagnosis of grade I varices, this study will define recurrent varices as the detection of grade II or III varices according to the modified Paquet classification (21).

The proportion of patients with recurrent varices and the corresponding 95% confidence interval (CI) will be calculated. Factors associated with recurrent varices will be compared between patients with and without recurrent varices. Continuous variables will be compared using the unpaired t test or Mann-Whitney U test as appropriate. For categorical variables, either the chi-square or Fisher exact test will be used. In the unlikely scenario where over 30 patients develop recurrent varices, a multivariable binary logistic regression model will be performed to identify independent factors associated with recurrent varices.

We hypothesise that non-invasive tests could detect recurrence of portal hypertension at earlier timepoints. Therefore, we will examine baseline and follow-up LSM, SSM, platelet count, and their combinations as potential predictors of recurrent varices.

#### 6.3 Secondary endpoints

#### Prevalence of varices in screening cohort

In the initial screening cohort of all patients who undergo endoscopy, we will calculate the proportion and 95% CI of patients with LSM <25 kPa who still harbour varices at baseline despite NSBB treatment and removal or suppression of the primary aetiological factor.

We will compare variables associated with varices between patients with and without varices at baseline. Continuous variables will be compared using unpaired t test or Mann-Whitney U test as appropriate, while categorical variables will be compared using the chi-square test or Fisher exact test. If over 30 patients exhibit varices at baseline, a multivariable binary logistic regression model will be performed to identify independent factors associated with varices.

#### Resumption of NSBB and variceal haemorrhage

For patients discontinuing NSBB, the secondary endpoint is resumption of NSBB or variceal haemorrhage during follow-up. The latter is defined as clinical symptoms of upper gastrointestinal bleeding (i.e., haematemesis, coffee ground vomiting, and/or tarry stool) and endoscopic evidence of variceal haemorrhage (active spurting or oozing from varices, or presence of stigmata of recent haemorrhage [e.g., red wale sign, cherry red spot, fibrin clot] with no alternative source of bleeding). The incidence rate of variceal haemorrhage, along with the 95% CI will be calculated. Factors associated with recurrent haemorrhage will be compared using the same statistical methods mentioned above. In the unlikely scenario where over 30 patients develop variceal haemorrhage, a multivariable Cox proportional hazard model will be applied to identify independent variables associated this event. Additionally, death and liver transplantation will be competing events precluding at-risk patients from developing variceal haemorrhage. Thus, should over 10% of the cohort either die or undergo liver transplantation during follow-up, a competing risk analysis will be conducted using the Fine-Gray model.

#### Other decompensating events

Other decompensating events include ascites and hepatic encephalopathy post-NSBB cessation, and the statistical methods used will be similar to those for variceal haemorrhage.

#### 6.4 Sample size calculation

In our previous study involving 818 patients with chronic hepatitis B and compensated advanced chronic liver disease well managed by oral antiviral drugs, only three (0.4%) developed variceal haemorrhage at a mean follow-up of 58 months (22). With a sample size of 300 patients, the study will have a two-sided 95% CI with a width of 0.037 (0.0125-0.0496) when up to 2.5% of patients develop the primary endpoint (23, 24). As per clinical practice standards, a miss rate of varices requiring treatment of up to 5% is generally considered acceptable for implementing non-invasive tests (10). Accordingly, this threshold (upper bound of the 95% CI <5%) will be taken as criteria of success (i.e., safe to discontinue NSBB according to the Baveno VII criteria). To mitigate the impact of potential patient dropout, we will allow for a dropout rate of up to 20%. Therefore, a total sample size of 375 patients is required.

#### 6.5 Anticipated challenges and contingency plans

Our team possesses the expertise and track records required to execute this study successfully. Our preliminary data support the feasibility of our sample size and event rate estimates. The study's multicentre design further bolsters the likelihood of its successful completion. In case of challenges in recruitment, we have plans to include additional collaborating sites. Currently, our university is leading a multicentre Asian study on the natural history of metabolic dysfunction-associated steatotic liver

disease with participating sites in China, Japan, South Korea, Taiwan, Malaysia and Singapore. There is potential to expand the proposed project and accelerate enrolment.

Given that this is the first prospective study examining the safety of NSBB discontinuation in this patient group, we will establish an independent Data and Safety Monitoring Board with planned interim analyses when the first 100 patients and all enrolled patients have reached 1 year of follow-up. If the rate of recurrent varices at 1 year exceeds 5% or if other safety concerns arise, the Board will recommend the study's early termination. In that case, Part 3 (NSBB-free follow-up for 10 years) would be discontinued. Patients with recurrent varices would resume NSBB, while those without recurrent varices or still within the first year of follow-up will be offered the options of resuming NSBB or regular endoscopic surveillance.

Endoscopy is an invasive procedure. Based on our previous clinical trials (25), a small percentage (typically <5%) of patients may decline the follow-up endoscopy at 1 year. These patients will still be included in the intention-to-treat and per protocol analyses as described above, ensuring that their data continues to contribute to the study's findings.

If a patient exhibits LSM <25 kPa at 1 year and refuses follow-up endoscopy, he/she will continue NSBB-free follow-up in Part 3 of this project, aligning with the Baveno VII recommendations. Conversely, if a patient exhibits LSM  $\geq$ 25 kPa at 1 year and declines the follow-up endoscopy, we will recommend resumption of NSBB.

#### 7. ETHICS

#### 7.1 Ethics review

The final study protocol, including the final version of the Informed Consent Form, must be approved in writing by the Joint The Chinese University of Hong Kong – New Territories East Cluster Clinical Research Ethics Committee (CUHK-NTEC CREC). The protocol must be re-approved by the CREC annually. All subsequent protocol amendments must be approved by the CREC.

#### 7.2 Ethical conduct of the study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/GCP, applicable regulatory requirements and the CREC.

#### 7.3 Informed consent

The investigator(s) will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study. The informed consent forms are

Stop-NSBB V1.0 dated 4 Dec 2023

available in traditional Chinese. Subjects must also be notified that they are free to discontinue from the

study at any time. The subject should be given the opportunity to ask questions and allow time to

consider the information provided. The subject's signed and dated informed consent must be obtained

before conducting any procedure specific for the study. The Principal Investigator must store the

original, signed Informed Consent Forms. One copy of the signed Informed Consent Form must be

given to the subject. If modifications are made according to local requirements, the new version has to

be approved by the CREC.

7.4 Data sharing

In line with current international standard of accountability and transparent reporting, data from this

study may be shared with outside parties upon reasonable request. Care will be taken to remove sensitive

data (name, identity numbers and dates of birth) before data sharing.

8. ADVERSE EVENT REPORTING

The adverse event reporting period for this study is from signing the informed consent through 6 months

of follow-up. Because the study will not involve study drugs or invasive procedures, there will not be

any per protocol post-treatment follow-up or adverse event reporting after the study period. Rather, an

appropriate clinic appointment will be arranged at the end of the study according to the clinical situation.

8.1 Adverse events

An adverse event is any undesirable medical event occurring in the subject within the trial period,

whether or not it is related to the study intervention.

The severity of an adverse event is defined as:

Mild: Transient symptoms, no interference with the subject's daily activities

--- J 1 )

Moderate: Marked symptoms, moderate interference with the subject's daily activities

Severe: Severe interference with the subject's daily activities.

The relationship of an adverse event to the study intervention is defined as:

Probable: Good reasons and sufficient documentation to assume a causal relationship

Possible: A causal relationship is conceivable and cannot be dismissed

Unlikely: The event is unlikely related to the study intervention

11

A telephone enquiry hotline for reporting subject's adverse events is available. The investigator will record all relevant information including signs and symptoms of the event, the onset time, the date of the event, the laboratory findings, concomitant drugs, and the outcome. All adverse events will be followed up until we have reached a defined outcome of the event, which can be one of the followings:

(1) recovered with sequelae (for chronic conditions), (2) recovered, or (3) the management of the adverse event is taken over by another physician when the study ends.

A clinical laboratory adverse event is any clinical laboratory abnormality that suggests a disease and/or organ toxicity is of sufficient severity that requires active intervention (i.e. change of dose, discontinuation of drug, more frequent follow-up or further investigation).

#### 8.2 Serious adverse events

A serious adverse event is an adverse event that results in one of the following outcomes:

- Death
- Life-threatening
- In-patient hospitalization or prolongation of existing hospitalization
- A persistent or significant disability or incapacity
- A congenital anomaly or birth defect

The definitions of causal relationship to study intervention are the same as those for adverse events. We have a 24-hour on-call system to handle serious adverse events. The investigator will assess and treat the subjects as soon as possible. A standard serious adverse event form will be used (provided by the CREC at <a href="http://intranet.ccter.cuhk.edu.hk/sae/">http://intranet.ccter.cuhk.edu.hk/sae/</a>) to report the events within 24 hours after acknowledgement. We will arrange unscheduled follow-up visits immediately or within 24 hours on receiving the subject's self-report of serious adverse events after the subjects have been discharged or if the subject has already been admitted to the hospital. Our investigators will assess the subject within 24 hours. The study team will record all relevant information including signs and symptoms of the event, the onset time, the date of the event, the laboratory findings, concomitant drugs, and the final outcome. A follow-up serious adverse event form will be sent within 14 days after submitting the initial serious adverse event form. Serious adverse events related to the study drug will be followed up until the subject has "recovered", "recovered with sequelae" or "died". SAE reports will be sent to our ethics committee. An unscheduled visit will be performed if subjects have to withdraw early from the study.

#### 9. REFERENCES

- 1. GBD Cirrhosis Collaborators. The global, regional, and national burden of cirrhosis by cause in 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Gastroenterol Hepatol 2020;5:245-66.
- 2. Villanueva C, Albillos A, Genesca J, Garcia-Pagan JC, Calleja JL, Aracil C, Banares R, Morillas RM, Poca M, Penas B, Augustin S, Abraldes JG, Alvarado E, Torres F, Bosch J. Beta blockers to prevent decompensation of cirrhosis in patients with clinically significant portal hypertension (PREDESCI): a randomised, double-blind, placebo-controlled, multicentre trial. Lancet 2019;393:1597-608.
- 3. Villanueva C, Torres F, Sarin SK, Shah HA, Tripathi D, Brujats A, Rodrigues SG, Bhardwaj A, Azam Z, Hayes PC, Jindal A, Abid S, Alvarado E, Bosch J, Carvedilol IPDMAg, the Baveno Cooperation: an EC. Carvedilol reduces the risk of decompensation and mortality in patients with compensated cirrhosis in a competing-risk meta-analysis. J Hepatol 2022;77:1014-25.
- 4. Liu KSH, Seto WK, Lau EHY, Wong DK, Lam YF, Cheung KS, Mak LY, Ko KL, To WP, Law MWK, Wu JT, Lai CL, Yuen MF. A Territorywide Prevalence Study on Blood-Borne and Enteric Viral Hepatitis in Hong Kong. J Infect Dis 2019;219:1924-33.
- 5. Wong VW, Wong GL, Woo J, Abrigo JM, Chan CK, Shu SS, Leung JK, Chim AM, Kong AP, Lui GC, Chan HL, Chu WC. Impact of the New Definition of Metabolic Associated Fatty Liver Disease on the Epidemiology of the Disease. Clin Gastroenterol Hepatol 2021;19:2161-71 e5.
- 6. Kwok R, Choi KC, Wong GL, Zhang Y, Chan HL, Luk AO, Shu SS, Chan AW, Yeung MW, Chan JC, Kong AP, Wong VW. Screening diabetic patients for non-alcoholic fatty liver disease with controlled attenuation parameter and liver stiffness measurements: a prospective cohort study. Gut 2016;65:1359-68.
- 7. Leung JC, Loong TC, Pang J, Wei JL, Wong VW. Invasive and non-invasive assessment of portal hypertension. Hepatol Int 2018;12:44-55.
- 8. Dajti E, Ravaioli F, Zykus R, Rautou PE, Elkrief L, Grgurevic I, Stefanescu H, Hirooka M, Fraquelli M, Rosselli M, Chang PEJ, Piscaglia F, Reiberger T, Llop E, Mueller S, Marasco G, Berzigotti A, Colli A, Festi D, Colecchia A, Spleen Stiffness IPDMASG. Accuracy of spleen stiffness measurement for the diagnosis of clinically significant portal hypertension in patients with compensated advanced chronic liver disease: a systematic review and individual patient data meta-analysis. Lancet Gastroenterol Hepatol 2023;8:816-28.
- 9. Kim HY, So YH, Kim W, Ahn DW, Jung YJ, Woo H, Kim D, Kim MY, Baik SK. Non-invasive response prediction in prophylactic carvedilol therapy for cirrhotic patients with esophageal varices. J Hepatol 2019;70:412-22.
- 10. de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C, Baveno VII Faculty. Baveno VII Renewing consensus in portal hypertension. J Hepatol 2022;76:959-74.
- 11. Wong GLH, Kwok R, Hui AJ, Tse YK, Ho KT, Lo AOS, Lam KLY, Chan HCH, Lui RA, Au KHD, Chan HLY, Wong VWS. A new screening strategy for varices by liver and spleen stiffness measurement (LSSM) in cirrhotic patients: A randomized trial. Liver Int 2018;38:636-44.
- 12. Wong GL, Liang LY, Kwok R, Hui AJ, Tse YK, Chan HL, Wong VW. Low Risk of Variceal Bleeding in Patients With Cirrhosis After Variceal Screening Stratified by Liver/Spleen Stiffness. Hepatology 2019;70:971-81.
- 13. Petta S, Sebastiani G, Bugianesi E, Vigano M, Wong VW, Berzigotti A, Fracanzani AL, Anstee QM, Marra F, Barbara M, Calvaruso V, Camma C, Di Marco V, Craxi A, de Ledinghen V. Non-invasive prediction of esophageal varices by stiffness and platelet in non-alcoholic fatty liver disease cirrhosis. J Hepatol 2018;69:878-85.
- 14. Wu CW, Lui RN, Wong VW, Yam TF, Yip TC, Liu K, Lai JC, Tse YK, Mok TS, Chan HL, Ng KK, Wong GL, Chan SL. Baveno VII Criteria Is an Accurate Risk Stratification Tool

- to Predict High-Risk Varices Requiring Intervention and Hepatic Events in Patients with Advanced Hepatocellular Carcinoma. Cancers (Basel) 2023;15.
- 15. Wu CW, Wong GL, Wong VW, Yam TF, Yip TC, Wong AC, Chan BW, Fong MM, Lai JC, Tse YK, Lee KF, Mok TS, Chan HL, Lui RN, Chan SL, Ng KK. Baveno VII criteria identify varices needing treatment in patients with hepatocellular carcinoma of different Barcelona Clinic Liver Cancer stages. J Gastroenterol Hepatol 2023;38:1381-8.
- 16. Lin H, Lai JC, Wong GL, Delamarre A, Ahn SH, Li G, Kim BK, Liang LY, Lee HW, Song SJ, Chan HL, Wong VW, de Ledinghen V, Kim SU, Yip TC. Risk and predictors of hepatic decompensation in grey zone patients by the Baveno VII criteria: A competing risk analysis. Aliment Pharmacol Ther 2023.
- 17. Marcellin P, Gane E, Buti M, Afdhal N, Sievert W, Jacobson IM, Washington MK, Germanidis G, Flaherty JF, Aguilar Schall R, Bornstein JD, Kitrinos KM, Subramanian GM, McHutchison JG, Heathcote EJ. Regression of cirrhosis during treatment with tenofovir disoproxil fumarate for chronic hepatitis B: a 5-year open-label follow-up study. Lancet 2013;381:468-75.
- 18. Lens S, Baiges A, Alvarado-Tapias E, E LL, Martinez J, Fortea JI, Ibanez-Samaniego L, Marino Z, Rodriguez-Tajes S, Gallego A, Banares R, Puente A, Albillos A, Calleja JL, Torras X, Hernandez-Gea V, Bosch J, Villanueva C, Garcia-Pagan JC, Forns X. Clinical outcome and hemodynamic changes following HCV eradication with oral antiviral therapy in patients with clinically significant portal hypertension. J Hepatol 2020;73:1415-24.
- 19. de Franchis R, Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol 2015;63:743-52.
- 20. Wong VW, Irles M, Wong GL, Shili S, Chan AW, Merrouche W, Shu SS, Foucher J, Le Bail B, Chan WK, Chan HL, de Ledinghen V. Unified interpretation of liver stiffness measurement by M and XL probes in non-alcoholic fatty liver disease. Gut 2019;68:2057-64.
- 21. Paquet KJ. Prophylactic endoscopic sclerosing treatment of the esophageal wall in varices -- a prospective controlled randomized trial. Endoscopy 1982;14:4-5.
- 22. Lee HW, Yip TC, Tse YK, Wong GL, Kim BK, Kim SU, Park JY, Kim DY, Chan HL, Ahn SH, Wong VW. Hepatic Decompensation in Cirrhotic Patients Receiving Antiviral Therapy for Chronic Hepatitis B. Clin Gastroenterol Hepatol 2021;19:1950-8 e7.
- 23. Brown LD, Cai TT, DasGupta A. Interval estimation for a binomial proportion. Stat Sci 2001;16:101-17.
- 24. Bland JM. The tyranny of power: is there a better way to calculate sample size? BMJ 2009;339:b3985.
- 25. Chan FKL, Ching JYL, Tse YK, Lam K, Wong GLH, Ng SC, Lee V, Au KWL, Cheong PK, Suen BY, Chan H, Kee KM, Lo A, Wong VWS, Wu JCY, Kyaw MH. Gastrointestinal safety of celecoxib versus naproxen in patients with cardiothrombotic diseases and arthritis after upper gastrointestinal bleeding (CONCERN): an industry-independent, double-blind, double-dummy, randomised trial. Lancet 2017;389:2375-82.